CLINICAL TRIAL: NCT00365339
Title: Randomized, Open-Label, Multiple-Dose Study to Evaluate the Effect of Famotidine on the Pharmacokinetics of Atazanavir/Ritonavir/Tenofovir in Healthy Subjects
Brief Title: Drug Interaction Study With Famotidine, Atazanavir, and Atazanavir/Ritonavir/Tenofovir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AI424-287
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections
Keywords: HIV; Protease Inhibitor
MeSH Terms: conditions — HIV Infections | interventions — Aripiprazole

ARMS (5):
- A (Active Comparator)
  Interventions: Drug: Atazanavir+Ritonavir+Tenofovir
- B (Experimental)
  Interventions: Drug: Atazanavir+Ritonavir+Tenofovir+Famotidine
- C (Experimental)
  Interventions: Drug: Atazanavir+Ritonavir+Tenofovir+Famotidine
- D (Experimental)
  Interventions: Drug: Atazanavir+Ritonavir+Tenofovir+Famotidine
- E (Experimental)
  Interventions: Drug: Atazanavir+Ritonavir+Tenofovir+Famotidine

INTERVENTIONS:
Drug: Atazanavir+Ritonavir+Tenofovir — Cap/Cap/Tablet, Oral, 300/100/300 mg, QAM/QAM/QAM, 10 days.
  Other Names: Abilify
  Arms: A
Drug: Atazanavir+Ritonavir+Tenofovir+Famotidine — Cap/Cap/Tablet/Tablet, Oral, 300/100/300/20 mg, QAM/QAM/QAM/Q12 coadmin, 7 days.
  Other Names: Abilify
  Arms: B
Drug: Atazanavir+Ritonavir+Tenofovir+Famotidine — Cap/Cap/Tablet/Tablet, Oral, 300/100/300/20 mg, QAM/QAM/QAM/Q12 2 hr post, 7 days.
  Other Names: Abilify
  Arms: C
Drug: Atazanavir+Ritonavir+Tenofovir+Famotidine — Cap/Cap/Tablet/Tablet, Oral, 300/100/300/40 mg, QAM/QAM/QAM/QPM 12 hr post, 7 days.
  Other Names: Abilify
  Arms: D
Drug: Atazanavir+Ritonavir+Tenofovir+Famotidine — Cap/Cap/Tablet/Tablet, Oral, 300/100/300/40 mg, QAM/QAM/QAM/Q12 2 hr post,7 days.
  Other Names: Abilify
  Arms: E

SUMMARY:
The purpose of this clinical research study is to assess the pharmacokinetics of atazanavir, identifying one or more dosing regimens of atazanavir/ritonavir/tenofovir when dosed with famotidine results in atazanavir exposures similar to those when atazanavir/ritonavir/tenofovir 300/100/300 mg is dosed without famotidine in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages 18 to 50 years old with a BMI 18 to 32 kg/m2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Assess PK of ATV, identifying dosing regimens of ATV/RTV/TDF when dosed with FAM that result in ATV exposures similar to ATV/RTV/TDF 300/100/300 mg with and without FAM.

SECONDARY OUTCOMES:
Assess PK , safety, and tolerability of ATV/RTV/TDF with and without FAM.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hamilton, New Jersey, United States